CLINICAL TRIAL: NCT06409286
Title: Assessment of Flow in Cerebrospinal Fluid Shunts With a Second Generation Wireless Thermal Anisotropy Measurement Device
Status: Not yet recruiting | Type: Observational
Sponsor: Rhaeos, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2024-01
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Hydrocephalus
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Shunted patients undergoing surgery: Patients with an existing implanted ventriculoperitoneal shunt who are experiencing shunt malfunction symptoms and require shunt revision surgery per standard of care shunt evaluation
  Interventions: Device: Thermal Anisotropy Measurement Device

INTERVENTIONS:
Device: Thermal Anisotropy Measurement Device — A wireless device for non-invasively assessing CSF shunt flow
  Other Names: FlowSense

SUMMARY:
This study evaluates the performance of a thermal anisotropy measurement device for non-invasively assessing CSF shunt flow. Patients with an existing implanted shunt and symptoms of shunt malfunction who require shunt revision surgery will be evaluated with the study device to assess flow in CSF shunts as confirmed by surgical outcomes at 7 days. If successful, this study will show that the study device accurately distinguishes between functioning (flowing) and non-functioning (non-flowing) shunts.

ELIGIBILITY:
Inclusion Criteria:

1. Existing ventriculoperitoneal CSF shunt on which the subject is dependent
2. At least one symptom of shunt malfunction as determined by the investigator, such as but not limited to seizure, fever, headache, vision problems, dizziness, disorientation, confusion, vomiting, lethargy, irritability, difficulty waking or staying awake, swelling along shunt tract, enlargement of head, loss of balance, gait disturbance, and loss of sensory or motor function
3. Exhibit shunt malfunction symptom(s) requiring surgical shunt revision per standard of care assessment without use of device data
4. Region of intact skin overlying an unambiguously identifiable chronically indwelling ventricular shunt which crosses the clavicle and is appropriate in size for application of the study device
5. Available for follow-up for up to seven days
6. Signed informed consent by subject or a parent, legal guardian, health care agent, or surrogate decision maker (according to local statutes, and collectively referred to as "surrogates" in this protocol)

Exclusion Criteria:

1. Presence of more than one distal shunt catheter in the study device measurement region
2. Presence of an interfering open wound or edema in the study device measurement area
3. Subject-reported history of adverse skin reactions to adhesives
4. Investigator judges that the subject is likely to be lost to follow-up due to unavailability or clinical outcome being unobtainable
5. Participation in the study will interfere with, or be detrimental to, administration of optimal health-care to the subject
6. Previous participation in a Rhaeos clinical study in which FlowSense device measurement data were acquired
7. Participation in any other investigational procedural, pharmaceutical, and/or device study that may influence the collection of valid data under this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric and adult shunt-dependent hydrocephalus patients with an existing ventriculoperitoneal (VP) shunt who are experiencing shunt malfunction symptoms and require shunt revision surgery per standard of care shunt evaluation without use of the study device data will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Flowsense Sensitivity | Upto 7 days
  The study device will yield an output of either "flow confirmed" or "flow not confirmed." Based on this assessment and the standard-of-care clinical treatment, each subject will fall into one of the following categories:
  True Positive (TP): Device outputs "flow not confirmed" AND a shunt revision surgery with confirmed shunt failure is performed False Positive (FP): Device outputs "flow not confirmed" AND either no shunt revision surgery is performed for 7 days or a shunt revision surgery without a confirmed shunt failure is performed True Negative (TN): Device outputs "flow confirmed" AND either no shunt revision surgery is performed for 7 days or a shunt revision surgery without a confirmed shunt failure is performed False Negative (FN): Device outputs "flow confirmed" AND a shunt revision surgery with confirmed shunt failure is performed
  Study device sensitivity will be calculated as TP / (TP + FN).

SECONDARY OUTCOMES:
Study device specificity, diagnostic accuracy, positive predictive value (PPV), negative predictive value (NPV), and diagnostic performance | Up to 7 days
  These secondary endpoints do not have associated success criteria. The study is not powered to achieve statistical significance for these endpoints.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States